CLINICAL TRIAL: NCT02237027
Title: Demonstration Project of Early Antiretroviral Therapy and Pre-exposure Prophylaxis for HIV Prevention Among Female Sex Workers in Cotonou, Benin
Brief Title: Early Antiretroviral Therapy and Pre-exposure Prophylaxis for HIV Prevention Among Female Sex Workers in Cotonou, Benin
Acronym: TasP/PrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Gilead Sciences (Industry); Imperial College London (Other); University of Bristol (Other); Johns Hopkins University (Other); Centre Muraz (Other); Université de Montréal (Other); Institut National en Santé Publique du Québec (Other); Université d'Abomey-Calavi (Other); National AIDS Control Organisation (Other)
Responsible Party: Principal Investigator, Michel Alary, Professor, MD, PhD, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPP1098973
Record Dates: First submitted 2014-08-20; First posted 2014-09-11 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2016-01

CONDITIONS: Adherence to Medication Regime
Keywords: HIV; Early treatment as prevention (TasP); Pre-exposure prophylaxis (PrEP); antiretroviral treatment; prevention; feasibility; female sex workers; Benin; West Africa
MeSH Terms: conditions — Medication Adherence | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TasP group (Experimental): HIV positive female sex workers receiving TasP using ART regimen as per Benin guidelines
  Interventions: Biological: TasP using ART regimen as per Benin guidelines
- PrEP group (Experimental): HIV negative female sex workers receiving PrEP using Truvada
  Interventions: Biological: PrEP using Truvada

INTERVENTIONS:
Biological: TasP using ART regimen as per Benin guidelines — Administration of ART to HIV positive female sew workers in order to prevent HIV transmission.
  Arms: TasP group
Biological: PrEP using Truvada — Administration of Truvada to HIV negative female sex workers in order to prevent HIV acquisition.
  Other Names: Combination of Tenofovir disoproxyl fumarate 300mg and Emtricitabine 200 mg
  Arms: PrEP group

SUMMARY:
In the last few years, early treatment of HIV-infected individuals, or "treatment as prevention (TasP), and pre-exposure prophylaxis with antiretroviral drugs among HIV-negative people at very high-risk of acquiring the infection (PrEP) have emerged as highly promising biological preventive interventions to tackle the HIV pandemic within the framework of combination prevention, a multi-component strategy that has been promoted for the last five years. In West Africa, the evidence strongly suggests that female sex workers (FSWs) contribute very disproportionally to the HIV spread. This is why the investigators propose this TasP and PrEP demonstration project in Benin, where our group has been involved in HIV prevention research in the sex work milieu for the last two decades.

After a run-in phase for community preparedness and the development of a specific education program on adherence, the investigators plan to recruit 100 HIV-infected FSWs in the TasP component of the project (these women will receive a first-line antiretroviral treatment (ART) regimen as per the Benin guidelines) and 250 HIV-negative FSWs in the PrEP component (these women will receive Truvada®). The recruitment period will last for one year, followed by an additional one year of follow-up, for a total follow-up period varying between 12 and 24 months, depending on when a given woman is recruited in the study. During follow-up visits every three months, the investigators will closely monitor treatment adherence and changes in sexual behaviour, including the use of viral load testing among TasP participants and Truvada® plasma level testing for PrEP participants, as well as detection of prostate-specific antigen (PSA) and Y-chromosome DNA in vaginal fluids in all participants.

The investigators will evaluate the feasibility of TasP and PrEP through a set of indicators, including uptake, coverage, adherence, condom migration, occurrence of side effects and development of drug resistance, whereas mathematical modeling will be used to predict the potential impact of both interventions in the sex work milieu and the general population, based on the actual set of indicators observed. The study will be completed by an economic evaluation of the interventions and a cost-effectiveness analysis.

Finally, the investigators will disseminate the results to the study population and to the Beninese health authorities and ensure the broad implementation of these interventions in Benin if the demonstration project shows that they are feasible and relevant.

DETAILED DESCRIPTION:
At the end of 2012, sub-Saharan Africa was home to 71% of the 35.3 million people living with HIV worldwide. Despite all the preventive and therapeutic efforts accomplished so far, the epidemic is persisting with approximately 1,600,000 new HIV infections occurring yearly in this region that is characterized by different epidemiological profiles. In West Africa, the epidemic is disproportionally concentrated among female sex workers (FSWs) who are involved directly or indirectly in 75% to 90% of HIV transmission cases towards the general population through "bridging" populations, essentially their clients and other male sexual partners. Hence, to achieve the control of the epidemic in this sub-region, especially in West Africa where the epidemic is much less generalized than in many other parts of the continent, it is important to tailor combination prevention including behavioural, structural, and biological components for the sex work milieu in general and FSWs in particular, in addition to ensuring adequate treatment of those already HIV-infected. However, despite substantial efforts in usual prevention methods in the last 10 years and effective reductions in the prevalence of HIV and other sexually transmitted infections (STIs) with concomitant increases in condom use in some countries, HIV prevalence is still high among FSWs in West Africa, with these highly vulnerable women having an HIV prevalence over 12 times higher than other women of reproductive age. Such a situation could constitute a threat to the progress achieved in controlling the HIV epidemic in this region.

Recently, in addition to previous preventive methods, such as consistent condom use and male circumcision, early treatment (treatment as prevention, TasP) has been shown to decrease HIV transmission by 96% in serodiscordant couples, whereas pre-exposure prophylaxis (PrEP) based on Tenofovir disoproxil fumarate or on the latter drug plus Emtricitabine (Truvada®) has been found to be 45 to 75% protective against HIV acquisition in four randomized controlled trials when used orally; no protection at all was observed in two trials conducted among women at high risk in African countries. These failures have now been shown to be mainly related to issues of poor adherence to the study drugs rather than poor biological efficacy. On the other hand, when combining data from several trials, the level of protection against HIV acquisition reached 90% among the sub-groups of trial participants achieving high levels of compliance. Based on the generally positive results obtained. Truvada® is now approved for PrEP by the Food and Drug Administration (FDA) in the USA. According to the Centers for Disease Control and Prevention, PrEP is largely considered a preventive individual-level intervention. However, it could potentially also have an impact at the population-level and help control the HIV epidemic if rolled out and adopted on a large scale for HIV prevention, especially among the most vulnerable populations. However, the feasibility of this approach is somewhat questioned by the low treatment adherence levels achieved in trials recruiting specifically highly vulnerable women in Africa. On the other hand, TasP can be viewed as a more classical public health intervention, as its population-level impact will largely depend on the coverage achieved in people at risk of transmitting HIV. However, the trial demonstrating TasP efficacy was carried out in serodiscordant couples, a population where treatment adherence may well be higher than in high-risk women who do not have a stable partner and who have shown lower levels of compliance than most other groups in the PrEP trials.

So far, antiretroviral therapy (ART) for all HIV-infected people, irrespective of their CD4 levels or clinical status (equivalent to TasP), is only recommended in the USA. However, the World Health Organization (WHO) and the United Nations Programme on HIV/AIDS (UNAIDS) have recently changed their recommendations on HIV treatment initiation of HIV positive individuals, increasing the eligibility criteria to treat when CD4 levels reach 500 cells/mm3 compared to the previously recommended threshold of CD4<350 cells/mm3. However, these changes have so far not been widely implemented at the country-level. Despite the proven efficacy of TasP and PrEP as prevention strategies in clinical trials, their efficiency must be evaluated in 'real life' situations, in various countries with specific cultural contexts, largely because the uptake of HIV testing, the acceptance of early treatment and PrEP as well as drug adherence may vary considerably according to personal, social and cultural characteristics, as clearly reflected by the variability in PrEP trial results. The absence of clear recommendations on both prevention strategies in different countries is partly due to the lack of evidence based on real world implementation especially amongst FSWs. The investigators are thus proposing this demonstration project among FSWs in Cotonou, Benin, to identify the best way to successfully implement TasP and PrEP in this specific setting. Benin is facing a concentrated epidemic with HIV prevalence estimated at 1.2% in a recent general population household survey, whereas HIV prevalence was estimated at 21% among FSWs in the latest integrated biological and behavioural survey (IBBS) carried out in 2012.

The project will use a field approach readily inserted within an ongoing combination prevention intervention, including clinical (for ex.: HIV testing and care, STI care) , behavioural (for ex.: non-governmental organization- and peer-led condom promotion) and structural components (for ex.: community empowerment, advocacy to decrease police harassment; community development activities leading to the constitution of FSW-led community based organizations), that the investigators implement in close collaboration with the National AIDS Control Programme (NACP) in most of the major cities and towns of Benin through a grant from the Canadian Institutes of Health Research (CIHR). The Dispensaire IST (DIST), a STI clinic dedicated to FSWs in Cotonou, will be the study clinic for this project.

TasP makes sense as a public health intervention as long as high levels of coverage are achieved in the high-frequency transmitter population targeted by this intervention. Hence, the TasP component of the project will benefit from the ongoing CIHR/NACP interventions aimed at increasing HIV testing among FSWs. Indeed, within this context, the investigators are currently carrying out a study on the determinants of regular HIV testing, based on the Theory of planned behaviour. The results of this study will be used to develop an education program promoting 3-monthly HIV testing among FSWs that will be ready to implement prior to the beginning of recruitment in the proposed study. The development of this program will use the intervention mapping approach. Its implementation is already planned in all the coverage area of our ongoing CIHR project. The latter project will also contribute by defining precise indicators of success specifically for professional FSWs (e.g. those whose main source of income is sex work who will constitute our target population), based on accurate estimations of their population size. Indeed, the investigators are currently conducting a detailed scientific mapping of the FSW population in the cities and towns covered by our ongoing intervention. The results of this size estimation study will be available before the end of 2013 and will be used to establish the denominators for the testing and TasP coverage indicators.

Contrary to TasP, PrEP is an individual preventive intervention for which the coverage level is of less importance. However, as the investigators are expecting that at least 60% of HIV-negative FSWs will accept PrEP, it may also have preventive benefits at the overall FSW population level. We have decided to combine TasP and PrEP in the same project for efficiency and ethical reasons. Indeed, this approach implies that all FSWs consulting at the project clinics will be offered some form of antiretroviral drugs with provision of adherence counseling. In addition, on an ethical point of view and considering the community perspective, it would be difficult to justify an approach where antiretroviral drugs would be given to HIV-negative women while asymptomatic HIV-positive FSWs with >350 CD4/mm³ are not treated. Note that according to the current Benin national guidelines, ART is provided for free to HIV-infected subjects with CD4<350 CD4/mm³, but this could change during the course of the study following the recently revised WHO guidelines proposing a threshold of 500 CD4/mm³ for treatment eligibility.

The proposed project is planned for three years: a 6-month phase-in period (submission of the project to all relevant ethics committees, community preparedness activities, conduction of a study on the determinants of the intention to adhere to ART regimens, for both HIV-positive and HIV-negative women, and development of an adherence education program based on theoretical frameworks and approaches similar to the ones used for the education program on regular testing mentioned above, development of study procedures), a 25-month follow-up period (including 12 months of active recruitment, and follow-up varying between 12 and 24 months) and a 5-month phase-out period to complete all the data entry, carry out the data analysis and disseminate the study results.

In the catchment area of the DIST, the investigators estimate that there are approximately 600 professional FSWs. Overall, the investigators are expecting to reach approximately 500 FSWs and to recruit and follow-up at least 90% of the HIV-positive (n~100) and at least 60% of the HIV-negative under PreP (n~250). Women eligible to ART under current guidelines and asymptomatic women with CD4 >350 cells/mm³ (TasP component) will be offered locally approved first line ART regimens while HIV-negative ones (PrEP component) will receive Truvada®. For all the analyses on TasP, the investigators will compare the women enrolled under the TasP component to those treated based on current national guidelines. Pregnant women and those still breastfeeding will be excluded from the PrEP component of the project. Women eligible to ART under current guidelines will receive their drugs through the NACP program, while those on TasP or PrEP will be supplied in drugs by this project.

In order to assess the potential impact of the combined TasP and PrEP interventions, the investigators will first compare the HIV incidence observed during the study to the 1.4 per 100 person-years incidence estimate from a follow-up study carried out among FSWs in Cotonou in the early 2010s. However, more importantly in terms of impact assessment, the investigators will use sophisticated carefully calibrated mathematical modelling techniques to estimate the impact of the intervention and each component on HIV transmission amongst FSWs, their clients and the general population, following modelling and impact assessment approaches previously developed for Cotonou and for the evaluation of Avahan, the India AIDS Initiative of the Bill & Melinda Gates Foundation.

Finally, the investigators will carry out prospective top down and patient level cost data collection mainly using a provider perspective approach, but also some patients perspective elements, and combine cost estimates with modeled impact projections in order to estimate the incremental cost-effectiveness of TasP and/or PrEP per HIV infection and disability adjusted life years (DALY) averted. Regression analysis will be used to determine if patient level costs are related to FSW characteristics (frequency of commercial sex, level of condom use, duration of sex work or age, and CD4 cell count at initiation of ART), ART provider or TasP/PrEP adherence and outcomes, and if deemed important these heterogeneities in the costs will be incorporated in modelling.

ELIGIBILITY:
TasP

* Inclusion Criteria:

  1. Being aged 18 years or more
  2. Being HIV-positive at screening and re-confirmed on a second sample
  3. Being HIV treatment naïve
* Exclusion Criteria:

  1. Women showing a compromised renal or liver function at clinical follow-up could be excluded anytime during the course of the study.

PrEP

* Inclusion Criteria:

  1. Being aged 18 years or more
  2. Being HIV-negative at screening and re-confirmed at the recruitment visit
* Exclusion Criteria:

  1. Being pregnant of breastfeeding
  2. Women showing a compromised renal or liver function at clinical follow-up could be excluded anytime during the course of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants adherent to treatment (self-report and pill count) | Change from day 14 to months 3, 6, 9, 12, 15, 18, 21 and 24
  To evaluate adherence to treatment in TasP and PrEP groups.
Percentage of participants adherent to treatment (drug dosage in plasma) | Change from day 14 to months 6, 12, and 24
  Quantification of tenofovir and emtricitabine in plasma to evaluate adherence to treatment in PrEP group.
Percentage of participants adherent to treatment (treatment failure) | Change from baseline to months 6, 12, 18, and 24
  Quantification of viral loads in TasP group to detect treatment failure, a very good marker of treatment adherence.

SECONDARY OUTCOMES:
Percentage of HIV seroconversion among participants from PrEP group | Change from baseline to months 3, 6, 9, 12, 15, 18, 21 and 24
  HIV testing to detect newly infected participants in order to evaluate PrEP efficiency in preventing HIV infection.
Occurence of side effects | Change from baseline to months 6, 12, 18, and 24
  Monitoring of complete blood count, glycaemia, renal function (creatinine level), and liver function (alanine aminotransferase level) to detect potential drug side effects in TasP and PrEP groups.
Change in condom use (self-report) | Change from baseline to months 3, 6, 9, 12, 15, 18, 21 and 24
  Self-report on condom use. To compare condom migration according to HIV status and treatment groups and detect a potential risk compensation.
Change in condom use (biomarkers) | Change from baseline to months 6, 12, and 24
  PSA and Yc-DNA, two biomarkers of unprotected intercourse, will be quantified in vaginal swabs to validate self-reported condom use in TasP and PrEP groups.
Development of drug resistance | Change from baseline to 24th month
  Genotyping of HIV in the TasP group at baseline and at 24 months in order to detect development of drug resistance to ART regimen.
Coverage of interventions | Baseline
  HIV testing coverage issues are critical for both TasP and PrEP feasibility so the proportion of the target population of professional FSWs who came for a screening visit will be assessed. The numerator of this indicator will be the number of people tested for HIV at screening and the denominator will be the number of professional sex workers in the catchment area of the study.
Uptake of PrEP intervention | Baseline
  Evaluation of the proportion of women enrolled in the PrEP group among FSWs testing HIV-negative at screening to determine if this preventive approach will be accepted as a useful addition to current protection practices adopted by HIV-negative FSWs.
Retention in the study | Change from baseline to every month until month 24
  Evaluation of the proportion of women that continue the study. The number of women eligible for each of follow-up visit will be used as the denominator at the moment when retention is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Alary, MD, PhD, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Dispensaire IST (DIST), Cotonou, Benin

REFERENCES:
- [Derived] Geidelberg L, Mitchell KM, Alary M, Mboup A, Behanzin L, Guedou F, Geraldo N, Goma-Matsetse E, Giguere K, Aza-Gnandji M, Kessou L, Diallo M, Keke RK, Bachabi M, Dramane K, Lafrance C, Affolabi D, Diabate S, Gagnon MP, Zannou DM, Gangbo F, Silhol R, Cianci F, Vickerman P, Boily MC. Mathematical Model Impact Analysis of a Real-Life Pre-exposure Prophylaxis and Treatment-As-Prevention Study Among Female Sex Workers in Cotonou, Benin. J Acquir Immune Defic Syndr. 2021 Feb 1;86(2):e28-e42. doi: 10.1097/QAI.0000000000002535. PMID 33105397